CLINICAL TRIAL: NCT05859308
Title: A Crossover Pilot Study of a Novel Virtual Reality Task in Parkinson's Disease Compared to a Group In-Person Rock Steady Boxing Program; Task Performance, Cognitive Outcomes, Perceptions, and Comparisons
Brief Title: A Novel Virtual Reality Task in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Amber Sousa, Assistant Professor, Neuropsychologist, New York Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1843
Record Dates: First submitted 2023-03-28; First posted 2023-05-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boxing (Active Comparator): Rock Steady Boxing
  Interventions: Other: Rock Steady Boxing
- Virtual Reality Pixel Plucker (Experimental): 30 minutes of VR engagement
  Interventions: Other: Virtual Reality Pixel Plucker

INTERVENTIONS:
Other: Virtual Reality Pixel Plucker — A virtual reality task where participants wear the Virtual Reality headset and respond to targets.
  Arms: Virtual Reality Pixel Plucker
Other: Rock Steady Boxing — An in-person boxing class designed for individuals with Parkinson's disease.
  Arms: Boxing

SUMMARY:
The purpose of this study is to compare experiences and effects of a virtual reality physical program to an in-person Rock Steady Boxing Program. People with Parkinson's disease, age 18 and up, who participate in Rock Steady Boxing weekly may join this study.

DETAILED DESCRIPTION:
If you agree to be in this study, we will ask you to do the following things:

Provide basic information about yourself, complete tests of thinking on the computer and in person, participate in your regular Rock Steady boxing, and for three weeks replace your Rock Steady Boxing with a virtual reality game done with a headset. You will work independently with a study team member.

* Visit 1 or Visit 1 and 2 if split up: Beginning Measures/Demographics, Parkinson's disease symptoms, Cognition (about 45 minutes), VR training (30 minutes) or Regular Rock Steady Boxing (1 hour)
* Visit 2-5: Virtual Reality training (30 minutes or Regular Rock Steady Boxing (1 hour)
* Visit 6: Virtual Reality training (30 minutes) or Regular Rock Steady Boxing (1 hour), Cognitive measures (about 20 minutes)
* Visit 7: Cognitive measures (about 20 minutes), Virtual Reality training (30 minutes) or Regular Rock Steady Boxing (1 hour); Intrinsic Motivation Inventory (5 minutes)
* Visit 8-11: Virtual Reality training (30 minutes) or Regular Rock Steady Boxing (1 hour)
* Visit 12 or Visit 13 if baseline was split up: Virtual Reality training (30 minutes) or Regular Rock Steady Boxing (1 hour), Cognitive Measures (20 minutes), Intrinsic Motivation Inventory (5 minutes), End of Study Survey (5-10 minutes)

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with Parkinson's disease
* Age 18+ years
* Currently involved in rock steady boxing
* Willing to participate 2-3 days/week

Exclusion criteria:

* Known history of movement-induced vertigo
* Other cognitive or movement disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Stroop Test, Inquisit Millisecond | through study completion, an average of one year
  measure of executive function

CONTACTS AND LOCATIONS:
Overall Officials: Amber Sousa, PhD, Principal Investigator — NYIT
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No